CLINICAL TRIAL: NCT03784261
Title: Usefulness of Non TNF Usage in Rheumatoid Arthritis Patients
Brief Title: Usefulness of Non TNF Usage in RA Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shinshu University (Other)
Responsible Party: Principal Investigator, Yukio Nakamura, Principle Investigator, Shinshu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NonTNF 2018
Record Dates: First submitted 2018-12-17; First posted 2018-12-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SAR, usually subucutaneous injection every 2 weeks (Active Comparator)
  Interventions: Drug: Drug: "Salirumab"; Drug: Drug: "Tocilizmab"; Drug: Drug: "Abatacept"
- TCZ, usually subucutaneous injection every 2 weeks (Active Comparator)
  Interventions: Drug: Drug: "Salirumab"; Drug: Drug: "Tocilizmab"; Drug: Drug: "Abatacept"
- ABT, usually subucutaneous injection every week (Active Comparator)
  Interventions: Drug: Drug: "Salirumab"; Drug: Drug: "Tocilizmab"; Drug: Drug: "Abatacept"

INTERVENTIONS:
Drug: Drug: "Salirumab" — To examine the effects of salirumab in RA patients
Drug: Drug: "Tocilizmab" — To examine the effects of tocilizmab in RA patients
Drug: Drug: "Abatacept" — To examine the effects of abatacept in RA patients

SUMMARY:
The aim of this study is to examine the efficacy and adverse events in the following 3 groups in rheumatoid arthritis patients:

1. Sarilumab treatment for 12 months
2. Tocilizmab treatment for 12 months
3. Abatacept treatment for 12 months

ELIGIBILITY:
Inclusion Criteria:

・RA patients

Exclusion Criteria:

* Not RA patients
* RA patients who are allergic to the drugs, refused to do this research, or who are pregnant

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-12-17 (Actual); Primary Completion 2022-12-16 (Estimated); Study Completion 2024-12-16 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Values of DAS28-CRP | Baseline and 1 year
  Assessment of efficacy in rheumatoid arthritis patients for 1 year treated by salirumab (N=30), tocilizumab (N=30), or abatacept (N=30).
Assessment of adverse event in rheumatoid arthritis patients for 1 year treated by salirumab (N=30), tocilizumab (N=30), or abatacept (N=30). | at 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Yukio Nakamura, Matsumoto, Nagano, Japan

IPD SHARING:
Plan to Share IPD: No